CLINICAL TRIAL: NCT01477671
Title: Prospective Dengue Seroprevalence Study in 5 to 10 Year-old Children in India
Brief Title: Prospective Dengue Seroprevalence Study in 5 to 10 Year-old Children
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DNG10; U1111-1124-7423 (Other: WHO)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue; Dengue Fever; Dengue Hemorrhagic Fever
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Participants aged between 5 and 10 year-old on day of inclusion.

SUMMARY:
This is a descriptive prospective community-based seroprevalence study.

Primary objective:

* To determine the prevalence of specific antibodies (immunoglobulin G [IgG]) against dengue in healthy 5 to 10 year-old children in India.

Secondary objectives:

* To determine the dengue virus serotype (DeNV-1,2,3 and /or 4) specific to the antibodies in positive (IgG) samples
* To estimate the prevalence of specific antibodies (IgG) against Japanese encephalitis in healthy 5 to 10 year-old children in India.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 5 and 10 year-old on the day of inclusion
* Healthy child as reported by the parent or legally qualified guardian
* Being registered in selected study site
* Provision of the informed consent form signed by at least one parent or legally qualified guardian
* For children between 8 and 10 years old, provision of the assent form signed.

Exclusion Criteria:

* N/A

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants aged between 5 and 10 year-old that are registered in health centers in India.
Sampling Method: Non-Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of positive samples with dengue specific serotype DENV 1, 2,3 and/or 4 | Baseline

SECONDARY OUTCOMES:
Prevalence of positive serum samples with JEV specific IgG antibodies | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (4):
- India (4):
  - Kalyani, West Bengali
  - Bangalore
  - Hyderabad
  - New Delhi

REFERENCES:
- [Result] Garg S, Chakravarti A, Singh R, Masthi NR, Goyal RC, Jammy GR, Ganguly E, Sharma N, Singh MM, Ferreira G, Moureau A, Ojha S, Nealon J; DNG10 study group. Dengue serotype-specific seroprevalence among 5- to 10-year-old children in India: a community-based cross-sectional study. Int J Infect Dis. 2017 Jan;54:25-30. doi: 10.1016/j.ijid.2016.10.030. Epub 2016 Nov 4. PMID 27825949
- [Derived] Bhavsar A, Tam CC, Garg S, Jammy GR, Taurel AF, Chong SN, Nealon J. Estimated dengue force of infection and burden of primary infections among Indian children. BMC Public Health. 2019 Aug 14;19(1):1116. doi: 10.1186/s12889-019-7432-7. PMID 31412836